CLINICAL TRIAL: NCT02768025
Title: Trial of Treatment Protocol for Smoking Cessation: A Pragmatic Randomized Controlled Pilot Study
Brief Title: Trial of Treatment Protocol for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daejeon University (Other)
Responsible Party: Principal Investigator, Sunju Park, Medical Doctor, Professor, Daejeon University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCKM_01
Record Dates: First submitted 2016-04-28; First posted 2016-05-11 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; tobacco control; acupuncture; Korean Medicine; Traditional & Complementary Medicine
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): NRT, counselling, traditional & complementary medicine treatment (Body acupuncture, Ear acupuncture and aromatic therapy).
  Interventions: Other: Traditional & Complementary Medicine treatment; Other: NRT, counselling
- Control group (Active Comparator): NRT, counselling
  Interventions: Other: NRT, counselling

INTERVENTIONS:
Other: Traditional & Complementary Medicine treatment — Body acupuncture, Ear acupuncture and aromatic therapy
  Arms: Intervention group
Other: NRT, counselling — Nicotine Replacement Therapy, counselling

SUMMARY:
Background: As smoking regulatory policies, including the WHO FCTC (Framework Convention on Tobacco Control), are enforcing, demand for smoking cessation treatment is being increased.

According the trend, development and evaluation of the medical guideline, Induced participation of medical personnel and available in Korean medical clinic, is needed. Purpose: To evaluate the satisfaction and effect of traditional & complementary medicine (T&CM) tobacco control program Methods: Recruited subjects were divided into control and test groups. They treated two times a week during the first three weeks and once a week during the last week.

Program participation rates and drop rates, satisfaction, amount of smoking before and after programs

, smoking-related key variables, nicotine dependence test (Fagerstrom test), Expired CO amounts, urinary cotinine amount, withdrawal symptoms, the change in quality of life(EQ-5D) are measured.

DETAILED DESCRIPTION:
Subjects in control group are treated NRT and counselling. Nicotine Replacement Therapy is provided 7 patches and 30 gums once a week for 4 weeks. Using amounts are depend on each subject's cravings. (Investigator will check how much they used.) Doctor consults about 10-15 minutes per visit.

Subjects in intervention group are treated NRT, counselling and traditional & complementary medicine treatment (Body acupuncture, Ear acupuncture and aromatic therapy). Body acupoints are HT7, LI4, ST36, LU7, LU6 on both sides. Ear acupoints are Shenmen, Lung, Pharynx, Trachea, Endocrine. Subjects are treated with acupuncture for 20 minutes per visit and put ear acupuncture like sticker for 1-2 days. Mixture oil of Lavender, peppermint, rosemary are used to massage behind the ears. It is used 2 times a day and they can adjust frequency depending on their cravings.(Investigator will check how much they used.)

ELIGIBILITY:
Inclusion Criteria:

* 1) having willing to stop smoking 2) currently smoking and applying one of the following

Exclusion Criteria:

* 1) suffering in the last 2 weeks cardiovascular disease or Severe arrhythmias, unstable angina 2) suffering from severe arrhythmia

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Continuous Abstinence Rate | 4 week
  endpoint of treatment

SECONDARY OUTCOMES:
7-day Point Prevalence Abstinence | 6,8,12,16,24 week
  follow-up measure
Prolonged Abstinence Rate | 3,6 month
  follow-up measure
Program participation rate | 0,7,10,14,17 day, 3,4,6,8,12,16,24 week
  each treatment and follow-up
Amount of smoking | 0,7,10,14,17 day, 3,4,6,8,12,16,24 week
  each treatment and follow-up
Tobacco craving | 0,7,10,14,17 day, 3,4,6,8,12,16,24 week
  each treatment and follow-up
Exhaled Carbon monoxide monoxide | 0,7,10,14,17 day, 3,4,6,8,12,16,24 week
  each treatment and follow-up
Quality of life | 0,4 week
  beginning and endpoint of treatment
Nicotine dependence test (Fagerstrom test) | 10, 17 day, 4week
Withdrawal symptoms | 1,2,3,4 week

CONTACTS AND LOCATIONS:
Overall Officials: Choong sik Cho, Doctor, Principal Investigator — Daejeon University
Locations (1):
- Dunsan Korean Medicine Hospital of Daejeon University, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No
This is confidential.

REFERENCES:
- [Derived] Jang S, Park S, Jang BH, Park YL, Lee JA, Cho CS, Go HY, Shin YC, Ko SG. Study protocol of a pragmatic, randomised controlled pilot trial: clinical effectiveness on smoking cessation of traditional and complementary medicine interventions, including acupuncture and aromatherapy, in combination with nicotine replacement therapy. BMJ Open. 2017 Jun 2;7(5):e014574. doi: 10.1136/bmjopen-2016-014574. PMID 28576892